CLINICAL TRIAL: NCT02152033
Title: Feasibility and Acceptability of Home-based Continuing Care
Brief Title: Home-based Continuing Care for Young Adults Leaving Residential Substance Abuse Treatment
Acronym: HCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Treatment Research Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: Public Health Management Corporation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R21DA036818 (NIH); R21DA036818 (NIH)
Record Dates: First submitted 2014-05-20; First posted 2014-06-02 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Substance Use Disorders
Keywords: Substance Abuse; Continuing Care; Recovery; Substance Abuse Treatment; Parent; Family; Young Adult
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home-based Continuing Care (Experimental): The components of Home-based Continuing Care (HCC) include brief parent training, brief Young Adult (YA) orientation and recovery planning, telephone-based continuing care (TCC) and home-based contingency management. Both parent and YA participants will attend sessions with a family specialist.
  Interventions: Behavioral: Home-based Continuing Care
- Services as Usual (Other): YAs completing residential care usually are referred to continuing outpatient services and/or self-help groups.
  Interventions: Behavioral: Services as Usual

INTERVENTIONS:
Behavioral: Home-based Continuing Care — All sessions will occur over the phone or Cisco WebEx meetings. Parents will participate in 5 individual sessions and 1 joint session with their child (45-50 min. each). Young Adults (YAs) will participate in 1-3 individual meetings (30- 45 min. each) and 1 joint session (45-50 min.). In addition, YAs will be contacted weekly for the first 8 weeks of HCC, then every other week for the remaining 24 weeks (20 calls total). He or she will be asked questions addressing risk and protective factors for relapse. Finally, parents will be trained to collect and test their child's urine sample and deliver incentives to the YA contingent upon biologically-verified abstinence and verified engagement in continuing service plan activities. Urine samples will be collected regularly over a 32 week period.
  Arms: Home-based Continuing Care
Behavioral: Services as Usual — Young Adults (YAs) will be told to follow the continuing service plan recommended by the residential treatment program. Parents will be told to support this and be sent information on continuing care developed by the Treatment Research Institute and the Partnership @ Drugfree.org (http://continuingcare.drugfree.org). We will provide no supplemental services during the study. We will train parents; however, on how to collect urine samples for research purposes only. They will not be trained on how to test the urine sample, only how to collect it and mail the sample to our staff for testing. We will offer separate 4 hour-workshops to parents and YAs after they have completed participation as an added study participation incentive for this group.
  Arms: Services as Usual

SUMMARY:
The purpose of this project is to develop and test a Home-based Continuing Care intervention that will help parents support the recovery of their Young Adult (YA) child who is leaving residential substance abuse treatment. The two phase pilot study will 1) interview 50 parents and 50 YAs recruited from residential treatment programs and from parent groups to inform the development of the intervention and 2) conduct a two-arm pilot study that will recruit a maximum of 20 parents and their young adult children into one of two conditions (Home-based Continuing Care [HCC] intervention group or Services as Usual [SAU] comparison group) with the main goal of determining whether conducting such an intervention is acceptable and sustainable, and to collect preliminary efficacy data. We hypothesize that pilot testing will indicate that: (a) HCC is acceptable and potentially sustainable; (b) conducting a randomized clinical trial is feasible, and (c) the magnitude of outcomes from HCC will be clinically meaningful.

DETAILED DESCRIPTION:
Several models of continuing care (CC) have been studied for adolescents and Young Adults (YAs) including online relapse prevention, brief telephone counseling and Assertive Continuing Care (ACC). Five sessions of in-person therapy or brief telephone counseling both have reduced relapse in youth completing treatment relative to a no CC condition, consistent with a growing body of research with adults supporting the efficacy of telephone-based CC (TCC). ACC has been thoroughly evaluated for adolescents. Some applications also have incorporated contingency management (CM) for engaging in activities including needed services; but ACC has not applied CM to biologically-verified abstinence -- an efficacious approach in adult CC. A significant drawback of ACC is that it is quite intensive, requiring extended clinician training and home visits. This increases the costs of the intervention and the difficulty of dissemination and implementation; therefore we plan to develop a less clinician-intensive continuing care model for YAs.

The two phase pilot study will 1) interview 50 parents and 50 YAs recruited from residential substance abuse treatment programs and from parent groups to inform the development of the intervention and 2) conduct a two-arm pilot study that will recruit a maximum of 20 parents and their YA children into one of two conditions (Home-based Continuing Care [HCC] intervention group or Services as Usual [SAU] comparison group) with the main goal of determining whether conducting such an intervention is acceptable and sustainable, and to collect preliminary efficacy data. We hypothesize that pilot testing will indicate that: (a) HCC is acceptable and potentially sustainable; (b) conducting a randomized clinical trial is feasible, and (c) the magnitude of outcomes from HCC will be clinically meaningful.

ELIGIBILITY:
Inclusion Criteria:

* Parent is 21 years of age or older
* Young Adult (YA) is 18-25 years of age
* YA's primary drug of abuse is prescription or other opiates
* Parent must be the custodial parent or former guardian or other caretaker of the YA
* YA is in residential treatment
* Parent and YA plan to live in the same residence during the intervention (32 weeks)
* Both Parent and YA provide written informed consent and pass the consent quiz testing knowledge of basic elements of informed consent and study requirements (including home urine testing).

Exclusion Criteria:

* Parent currently has a substance use disorder (SUD) as determined via DSM-IV-TR criteria or a history of SUD and in recovery for less than 2 years
* Parent or YA has been diagnosed as having, or behaves in, a manner consistent with having significant cognitive impairment (e.g., an unrelieved psychosis or other serious mental illness)
* YA reports suicidal ideation with a plan, or engaged in suicidal behavior during residential treatment
* YA has a recent history of severe violence toward the parent (e.g., involving weapons or hospitalization)
* YA's residential program provides comprehensive continuing services
* YA does not consent to participation within 2 weeks of discharge

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in Young Adult Drug Use from Baseline to 16 week and 32 week follow-ups | Baseline, Weekly, 16 week and 32 week follow-ups
  Young Adult participants will complete a Timeline Follow Back (Baseline, 16 week and 32 week follow-ups) and provide a urine sample to be tested for drug and alcohol use (Baseline, Weekly, 16 week and 32 week follow-ups).

SECONDARY OUTCOMES:
Change in Parent and Young Adult Relationship Satisfaction from Baseline to 16 week and 32 week follow-ups | Baseline, 16 week and 32 week follow-ups
  Parent participants will complete the Parent Happiness with Youth Scale and young adult participants will complete the Youth Happiness with Parents scale.
Parent and Young Adult Treatment Retention | 32 weeks post baseline
  Weeks of participation in the home-based continuing care intervention
Parent and Young Adult Recruitment Rate by percent approached | 10 month recruitment period
  We will measure the percent of young adults and parents that were approached and agreed to participate in the study.
Parent and Young Adult Engagement in HCC by urine sample collected | 32 week intervention period
  We will measure the percent of urine samples the parent collects from the young adult.
Parent and Young Adult Treatment Acceptability | 16 week and 32 week follow-ups
  Participants will complete the Treatment Evaluation Inventory
Parent and Young Adult Research Retention | 16 week and 32 week follow-ups
  Follow-up rates
Parent and Young Adult Engagement in HCC by number of calls completed | 32 week intervention period
  We will measure the number of telephone counseling calls completed by the parent and young adult.
Parent and Young Adult Recruitment Rate by monthly recruitment rate | 10 month recruitment period
  We will measure the mean number of parent and young adult participants that are recruited per month.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly C Kirby, Ph.D., Principal Investigator — Treatment Research Institute
Locations (1):
- Family Training Program, Philadelphia, Pennsylvania, United States